CLINICAL TRIAL: NCT04297007
Title: Comparison of Ultrasound-Guided Type-II Pectoral Nerve Block and Rhomboid Intercostal Block for Pain Management Following Mastectomy Surgery
Brief Title: Pectoral Nerve Block Type-II and Rhomboid Intercostal Block for Pain Management Following Mastectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol Hospital 9
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Diseases; Breast Fibroadenoma
Keywords: Mastectomy and axillary dissection surgery; Pectoral nerve block; Rhomboid intercostal block; Postoperative pain management
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Fibroadenoma

STUDY DESIGN:
Intervention Model Description: There are three models for this study. Patients will be randomly divided into three groups (Group P = PECS group, Group R = RIB group, Group C = Control group), before entering the operating room.
Who Masked: Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group P = PECS-II group (Active Comparator): In group P, PECS will be performed with patients in the supine position at the end of the surgery before extubation by using US (Vivid Q, GE Healthcare, US). Under aseptic conditions the high frequency linear probe (11-12 MHz) will be covered with a sterile sheath and a 22G, 50 mm block needle will be used. US probe will be placed on the 4th rib. The muscles PMm, Pmm and Sam will be visualized. At the anterior axillary level or mid-axillary level, via the in-plane technique, Pecs II will be applied by injecting 20 mL of 0.25% bupivacaine in a cephalad to caudad direction to the fascia on Sam.
  Interventions: Other: PECS block
- Group R = RIB group (Active Comparator): In group R, RIB block will be performed with patients in the lateral decubitus position at the end of the surgery before extubation. The linear high frequency probe will be placed in sagittal plane medially on the medial border of the scapula at T5-6 level. The trapezius muscle, rhomboid major muscle, intercostal muscle, ribs and the pleura will be visualized. The needle will be inserted into the fascial plane between the rhomboid major and intercostal muscles in a cranio-caudal direction. A dose of 20 ml 0,25% bupivacaine will be injectted into the fascial plane.
  Interventions: Other: Rhomboid intercostal block
- Group C = Control group (No Intervention): A dose of ibuprofen 400 mgr and tramodol 100 mg will be performed intraoperatively. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.

INTERVENTIONS:
Other: PECS block — A dose of ibuprofen 400 mgr and tramodol 100 mg will be performed intraoperatively. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.
  Arms: Group P = PECS-II group
Other: Rhomboid intercostal block — A dose of ibuprofen 400 mgr and tramodol 100 mg will be performed intraoperatively. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit.
  Arms: Group R = RIB group

SUMMARY:
Postoperative pain is an important issue in patients underwent mastectomy and axillary dissection surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay. The US-guided pectoral nerve block (PECS) may be used for postoperative pain treatment following breast surgery. It is a novel interfascial block that was defined by Blanco. Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. Local anesthetic solution is administrated between the rhomboid muscle and intercostal muscles over the T5-6 ribs. It has been reported that RIB may provide effective analgesia management for several breast surgeries.

The primary aim of the study is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Postoperative pain is an important issue in patients underwent mastectomy and axillary dissection surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following mastectomy and axillary dissection surgery. Ultrasound (US)-guided interfascial plane blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. The US-guided pectoral nerve block (PECS) may be used for postoperative pain treatment following breast surgery. It is a novel interfascial block that was defined by Blanco. It is easy to perform; under ultrasound (US) guidance, the interfascial region between the pectoral muscles (pectoralis major (PMm) and minor (Pmm), serratus anterior Sam) is injected with local anaesthetics. It has been reported that PECS type-2 block provides effective analgesia management for mastectomy and axillary dissection surgeries.

Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. Local anesthetic solution is administrated between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2-3 cm medially of the medial border of the scapula. RIB targets both the posterior rami and lateral cutaneous branches of the thoracic nerves and provides analgesia for the hemithorax from T2 to T9. It has been reported that RIB may provide effective analgesia management for several breast surgeries.

The aim of this study is to evaluate the efficacy of the US-guided PECS-II and RIB for postoperative analgesia management compare to no intervention control group after mastectomy and axillary dissection surgery. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for mastectomy and axillary dissection surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Karaca O, Pinar HU, Arpaci E, Dogan R, Cok OY, Ahiskalioglu A. The efficacy of ultrasound-guided type-I and type-II pectoral nerve blocks for postoperative analgesia after breast augmentation: A prospective, randomised study. Anaesth Crit Care Pain Med. 2019 Feb;38(1):47-52. doi: 10.1016/j.accpm.2018.03.009. Epub 2018 Apr 5. PMID 29627431
- [Background] Tulgar S, Selvi O, Thomas DT, Manukyan M, Ozer Z. Rhomboid intercostal block in a modified radical mastectomy and axillary curettage patient; A new indication for novel interfascial block. J Clin Anesth. 2019 May;54:158-159. doi: 10.1016/j.jclinane.2018.12.006. Epub 2018 Dec 13. No abstract available. PMID 30553225